CLINICAL TRIAL: NCT01358253
Title: Prospective Study of Rituximab Combined With Chemotherapy for CD20+ Adult Acute Lymphoblastic Leukemia
Brief Title: Rituximab Plus Chemotherapy for CD20+ Adult Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Zhao Weili/Professor, Department of hematology Ruijin Hospital/Shanghai Institute of hematology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ-2010-56
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Rituximab; HyperCVAD
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Dexamethasone; Cytarabine; Methotrexate; Rituximab; Mercaptopurine; Prednisone; Asparaginase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HyperCVAD (Active Comparator): Consolidation:
  HyperCVAD(odd courses) alternated with high-dose methotrexate + cytarabine (even courses) every 21 days or later to allow for myelosuppression recovery, for total of 8 courses.
  Maintenance:
  6-Mercaptopurine+Methotrexate for 24 months. Vincristine+Prednisone for the first 12 months. L-asparaginase in month 3 and 9.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Dexamethasone; Drug: Cytarabine; Drug: Methotrexate; Drug: 6-Mercaptopurine; Drug: Prednisone; Drug: L-asparaginase
- R-HyperCVAD (Experimental): Consolidation:
  R-HyperCVAD(odd courses) alternated with high-dose methotrexate + cytarabine (even courses) every 21 days or later to allow for myelosuppression recovery, for total of 8 courses.
  Maintenance:
  6-Mercaptopurine+Methotrexate for 24 months. Vincristine+Prednisone for the first 12 months. L-asparaginase in month 3 and 9. Rituximab in month 6 and 12.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Dexamethasone; Drug: Cytarabine; Drug: Methotrexate; Drug: Rituximab; Drug: 6-Mercaptopurine; Drug: Prednisone; Drug: L-asparaginase

INTERVENTIONS:
Drug: Cyclophosphamide — 300 mg/m2 IV over 3 hours every 12 hours x 6 doses days 1, 2, 3 (total dose 1800 mg/m2)(odd courses).
Drug: Doxorubicin — 50 mg/m2 IV over 2-24 hours via CVC on day 4 after last dose of cyclophosphamide given (odd courses).
Drug: Vincristine — Consolidation:1.4 mg/m2 (max 2mg) IV on day 4 and day 11 (odd courses). Maintenance:1.4mg/m2(max 2mg) IV monthly from 1st to 12th month.
Drug: Dexamethasone — 40mg IV or by mouth (P.O.) daily days 1-4 and days 11-14(odd courses)
Drug: Cytarabine — 2g/m2 IV over 2 hours every 12 hours for 4 doses on days 2, 3 (even courses).
Drug: Methotrexate — Consolidation:1000 mg/m2 IV over 24 hours on day 1 (even courses). Maintenance:25mg/m2 weekly for 24 months.
Drug: Rituximab — Consolidation:375 mg/m2 IV day 1 for the odd courses of therapy (total 4 times).
  Maintenance:375 mg/m2 IV in 6th month and 12th month.
  Arms: R-HyperCVAD
Drug: 6-Mercaptopurine — Maintenance:60mg/m2 daily for 24 months.
Drug: Prednisone — Maintenance:40mg/m2 from days 1-7 monthly from 1st to 12th month.
Drug: L-asparaginase — Maintenance:6000IU/m2 IV on days 1,3,5 of the 3rd and 9th month.

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of Rituximab combined with chemotherapy in CD20+ adult acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is a group of biologically heterogeneous diseases with diverse prognosis. Novel strategies for adult ALL have approached a CR rate of over 80%, which is similar to pediatric ALL. But the long term survival of adult ALL is only 30%-40%, much lower than pediatric patients.

In our trial, all the patients will first receive Vincristine 1.4mg/m2, max 2mg IV days 1,8,15,22, Daunorubicin 45mg/m2 IV days 1-3,Cyclophosphamide 750mg/m2 IV day 1 and prednisone 40-60mg/m2,by mouth days 1-14 (VDCP)regimen as initial induction therapy. If patients achieve complete remission after induction, they will be enrolled in our study for further consolidation and maintenance. If the tumor cells in bone marrow remain 5% to 20% after induction, the patients will receive VDCLP(VDCP+L-asparaginase 6000IU/m2 IV days5,7,9,11,13) and be enrolled until complete remission.

Rituximab is the main experimental intervention in our study.The consolidation regimen is HyperCVAD/MA or R-HyperCVAD/MA for totally 8 courses. The maintenance regimen includes 6-Mercaptopurine+Methotrexate for 24 months, Vincristine+Prednisone for the first 12 months, L-asparaginase in month 3 and 9 with or without Rituximab in month 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD20-positive ALL
* Adequate liver function (bilirubin less than or equal to 1.5*ULN, unless considered due to tumor), and renal function (creatinine less than or equal to 1.5*ULN, unless considered due to tumor)
* Signed informed consent

Exclusion Criteria:

* Prior history of treatment with high-dose Ara-C, MTX or rituximab
* Pregnant or lactating women
* History of allergy to rituximab
* Unable to sign informed consent
* Active replication of HBV
* History of stem cell transplantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
CR duration | After two 21-day courses
  Bone marrow MRD examination every two months
disease free survival | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, MD,PhD, Principal Investigator — Department of hematology Ruijin Hospital/Shanghai Institute of Hematology
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China